CLINICAL TRIAL: NCT00590226
Title: Comparative Trial Between Insulin Detemir Versus NPH Insulin In Hospitalized Patients With Type 2 Diabetes
Brief Title: Insulin Detemir Versus NPH Insulin In Hospitalized Patients With Diabetes
Acronym: DEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00048954; 791-2006 (Other: Other)
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; inpatient hyperglycemia; SQ insulin; Hospitalized patients with type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart; Insulin, Isophane; Insulin; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- detremir + aspart insulin (Experimental): Detemir insulin once daily + aspart insulin before meals three times a day at an initial total dose of 0.5 units/kg/day, subcutaneously
  Interventions: Drug: Detemir + aspart insulin before meals
- NPH + regular insulin (Active Comparator): NPH insulin once a day + regular insulin before breakfast and dinner at an initial total dose of 0.5 units/kg/day, subcutaneously
  Interventions: Drug: NPH insulin + regular insulin

INTERVENTIONS:
Drug: Detemir + aspart insulin before meals — Detemir insulin SQ once daily + aspart insulin SQ before meals
  Other Names: levemir; novolog
  Arms: detremir + aspart insulin
Drug: NPH insulin + regular insulin — NPH insulin SQ + regular insulin SQ before breakfast and dinner
  Other Names: novolin N; novolin R
  Arms: NPH + regular insulin

SUMMARY:
High blood glucose levels in hospitalized patients with diabetes are associated with increased risk of medical complications. Improved glucose control with insulin injections may improve clinical outcome and prevent some of the hospital complications. It is not known; however, what is the best insulin regimen in hospitalized patients. Recently, the use of basal/bolus insulin therapy with detemir (Levemir®) and rapid-acting insulin (lispro, aspart, glulisine) has been shown to facilitate outpatient glycemic control with lower rate of hypoglycemic (low blood sugar) events in patients with diabetes. In this study, we will determine the efficacy and safety of the combination of detemir and aspart insulin in the inpatient management of subjects with diabetes. We hypothesize that in patients with type 2 diabetes admitted to general medicine wards, treatment with insulin detemir once daily plus insulin aspart before meals will allow better glycemic control and lower rate of hypoglycemic events than treatment with twice a day NPH plus regular insulin before meals. Detemir is a long-acting insulin which is given subcutaneously (under the skin) once daily. Aspart is a rapid-acting insulin which is given subcutaneously several times a day and frequently before meals. Detemir and aspart insulins are approved for use in the treatment of patients with diabetes by the FDA.

This investigator-initiated research will be conducted at Grady Memorial Hospital, Atlanta and at Rush University Medical Center, Chicago, IL. Dr. Umpierrez designed the study and will serve as principal investigator. A total of 65 patients will be recruited at Grady and 65 patients at the Rush University Medical Center, Chicago, IL.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 70 years admitted to a general medical service.
2. A known history of type 2 diabetes mellitus > 3 months, receiving any combination of oral antidiabetic agents (sulfonylureas, metformin, thiazolidinediones) and/or insulin therapy.
3. Subjects must have an admission blood glucose > 140 mg and < 400 mg/dL and no evidence of ketoacidosis (serum bicarbonate < 18 mEq/L, venous or arterial pH < 7.30, positive serum or urinary ketones).

Exclusion Criteria:

1. Subjects with increased blood glucose concentration, but without a known history of diabetes.
2. Subjects with a history of acute hyperglycemic crises such as diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria [63].
3. Patients with acute critical or surgical illness and/or expected to require admission to a critical care unit (ICU, CCU), or to undergo surgery during the hospitalization course.
4. Patients with clinically relevant hepatic disease (ALT 2.5x > upper limit of normal), or impaired renal function, as shown by a serum creatinine ≥2.0 mg/dL for males, or ≥ 1.8 mg/dL for females.
5. History of drug or alcohol abuse within the last 2 years.
6. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
7. Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, such as hypercortisolism, acromegaly, or hyperthyroidism.
8. Female subjects are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Baldwin, MD, Study Chair — Rush University Medical Center
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois

REFERENCES:
- [Result] Umpierrez GE, Hor T, Smiley D, Temponi A, Umpierrez D, Ceron M, Munoz C, Newton C, Peng L, Baldwin D. Comparison of inpatient insulin regimens with detemir plus aspart versus neutral protamine hagedorn plus regular in medical patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):564-9. doi: 10.1210/jc.2008-1441. Epub 2008 Nov 18. PMID 19017758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Grady Memorial Hospital in Atlanta, GA and at Rush University Medical Center, Chicago, IL. IRB approval was given at each center and consent was obtained from all subjects. Patients with a h/o T2DM were recruited in 2007.
Groups:
- Detemir + Aspart: Detemir insulin once daily + aspart insulin before meals
- NPH+Regular: NPH insulin + regular insulin before breakfast and dinner
Period: Overall Study
Arm/Group | Detemir + Aspart | NPH+Regular
Started | 67 | 63
Completed | 67 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Detemir + Aspart | NPH+Regular | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 57 | 117
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10) | 58 (10) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  United States | 67 | 63 | 130

OUTCOME MEASURES:

1. Primary Outcome: Mean AM BG (mg/dl)
Description: average AM daily BG with detemir insulin once daily plus insulin aspart before meals and NPH insulin twice daily plus regular insulin before meals in patients with DM2
Time Frame: during hospitalization
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Detemir + Aspart | NPH+Regular
Number analyzed (Participants) | 67 | 63
mg/dl | 144 (56) | 155 (62)

2. Secondary Outcome: Number of Patients With Hypoglycemic Events
Description: number of patients with hypoglycemic events as defined as BG 40-59 mg/dl
Time Frame: during hospitalization
Measure: Number; unit: participants
Arm/Group | Detemir + Aspart | NPH+Regular
Number analyzed (Participants) | 67 | 63
participants | 15 | 13

ADVERSE EVENTS:
Time Frame: during study period in the hospital
Description: Hypoglycemic event is defined as blood glucose < 60 mg/dl. All serious adverse events were monitored.
Arm/Group | Detemir + Aspart | NPH+Regular
Serious Adverse Events (participants affected / at risk) | 15/67 | 13/63
Other Adverse Events (participants affected / at risk) | 0/67 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Detemir + Aspart (N=67) | NPH+Regular (N=63)
Hypoglycemia (Metabolism and nutrition disorders) | 15 (15) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No